CLINICAL TRIAL: NCT05866315
Title: The Effect of Remimazolam on Remifentanil-induced Hyperalgesia
Brief Title: The Effect of Remimazolam on Opioid Induced Hyperalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Wonkwang UH13
Record Dates: First submitted 2023-03-28; First posted 2023-05-19 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Hyperalgesia, Mechanical
Keywords: remifentanil; remimazolam; opioid-induced hyperalgesia
MeSH Terms: conditions — Hyperalgesia | interventions — remimazolam; Desflurane; Remifentanil

STUDY DESIGN:
Intervention Model Description: 1. Group RHR (Remimazolam- High doses of Remifentanil): Administer remimazolam at a dose of 6 mg/kg/h initially, followed by 1 mg/kg/h, and remifentanil at 0.3 µg/kg/min.
  2. Group DHR (Desflurane-High doses of Remifentanil): Administer desflurane at 1 MAC, adjusting the dose by 1 vol% titration to maintain MAP and BIS levels, and remifentanil at 0.3 µg/kg/min.
  3. Group DLR (Desflurane-Low-dose of Remifentanil): Administer desflurane at 1 MAC, adjust the dose by 1 vol% titration to maintain MAP and BIS levels, and remifentanil at 0.025 µg/kg/min.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A trained anesthesiologist not involved in general anesthesia assessed clinically relevant and mechanically evoked pain using the Von-Frey filaments and secondary outcomes after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group DLR (Active Comparator): Administer desflurane at 1 MAC, adjust the dose by 1 vol% titration to maintain MAP and BIS levels, and remifentanil at 0.025 µg/kg/min.
  Interventions: Drug: Desflurane; Drug: Remifentanil
- Group DHR (Experimental): Administer desflurane at 1 MAC, adjusting the dose by 1 vol% titration to maintain MAP and BIS levels, and remifentanil at 0.3 µg/kg/min.
  Interventions: Drug: Desflurane; Drug: Remifentanil
- Group RHR (Experimental): Administer remimazolam at a dose of 6 mg/kg/h initially, followed by 1 mg/kg/h, and remifentanil at 0.3 µg/kg/min.
  Interventions: Drug: Remimazolam; Drug: Remifentanil

INTERVENTIONS:
Drug: Remimazolam — Administer remimazolam
  Other Names: Byfavo
  Arms: Group RHR
Drug: Desflurane — administer desflurane
  Other Names: desfuralne
  Arms: Group DHR; Group DLR
Drug: Remifentanil — administer remifentanil
  Other Names: Ulitva

SUMMARY:
The goal of this prospective, randomized, controlled study is to investigate the effect of remimazolam on opioid-induced hyperalgesia (OIH) in patients undergoing single port-laparoscopically assisted urologic surgery.

The main question[s] it aims to answer are:

* [The mechanical hyperalgesia threshold]
* [Area of hyperalgesia around the surgical incision 24 h after surgery (cm^2)]

In three groups: Group RHR (Remimazolam- High-dose Remifentanil), Group DHR (Desflurane-low-dose Remifentanil) or Group DLR (Control).

DETAILED DESCRIPTION:
Ninety-three (n = 31 per group) American Society of Anesthesiologists I-II patients (age 20-65 years) will be scheduled for single port-laparoscopically assisted urologic surgery.

Group RHR (Remimazolam-Remifentanil): Administer remimazolam at a dose of 6 mg/kg/h initially, followed by 1 mg/kg/h, and remifentanil at 0.3 µg/kg/min.

Group DHR (Desflurane-Remifentanil): Administer desflurane at 1 minimum alveolar concentration (MAC), adjusting the dose by 1 vol% titration to maintain MAP and BIS levels, and remifentanil at 0.3 µg/kg/min.

Group DLR (Control): Administer desflurane at 1 MAC, adjust the dose by 1 vol% titration to maintain mean arterial pressure (MAP) and bispectral index (BIS) levels, and remifentanil at 0.3 µg/kg/min.

Mechanical hyperalgesia threshold, Time to first postoperative analgesic requirement (min), Injected PCA volume containing morphine for 12 h after surgery (ml), Pain intensity: VAS 1 h after surgery, VAS 6 h after surgery, VAS 12 h after surgery VAS 24 h after surgery. Area of hyperalgesia around the surgical incision 24 h after surgery (cm^2) will be checked.

ELIGIBILITY:
1. Inclusion criteria will include as follows; ASA(American Society of Anesthesiologists)physical status 1-2 patients, Age with 20-65 years, and Single port-laparoscopically assisted urologic surgery.
2. Exclusion criteria will include as follows; a known allergy to remimazolam or remifentanil, a history of drug or alcohol abuse, psychiatric disorders, acute cardiovascular disorders, or unstable hypertension, and other respiratory or neuromuscular pathology, treated with opioid-containing any analgesic drug within 24 h before surgery and contraindications to the self-administration of opioids (i.e., were unable to understand the PCA device).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
The mechanical hyperalgesia threshold | at 24 hours after surgery
  The mechanical hyperalgesia threshold (g/mm^2) (preoperative) and 2 cm from the single port incision site (postoperative) at four points (horizontally and perpendicularly).

SECONDARY OUTCOMES:
Time to first postoperative analgesic requirement | Within 1 hour after surgery
  Time to first postoperative analgesic requirement (min)
Injected PCA volume containing morphine for 24 h after surgery | 24 hours after surgery
  Injected PCA volume containing morphine for 24 h after surgery (ml)
Pain intensity | 1 hour after surgery
  The Visual analogue scales (VAS)-100 is a line with words describing the extremes of pain from "no pain" to "worst imaginable pain".
Pain intensity | 6 hours after surgery
  The Visual analogue scales (VAS)-100 is a line with words describing the extremes of pain from "no pain" to "worst imaginable pain".
Pain intensity | 12 hours after surgery
  The Visual analogue scales (VAS)-100 is a line with words describing the extremes of pain from "no pain" to "worst imaginable pain".
Pain intensity | 24 hours after surgery
  The Visual analogue scales (VAS)-100 is a line with words describing the extremes of pain from "no pain" to "worst imaginable pain".
Area of hyperalgesia around surgical incision | 24 hours after surgery
  Area of hyperalgesia around surgical incision (cm^2)

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Lee, M.D.,Ph.D., Study Director — Wonkwang University Hospital
Locations (2):
- South Korea (2):
  - Wonkwag UH, Iksan, Jeollabukdo
  - Wonkwang University hospital, Iksan

IPD SHARING:
Plan to Share IPD: No